CLINICAL TRIAL: NCT00447603
Title: A Randomized, Double-Blind, Active Comparator Study to Evaluate the Antihypertensive Efficacy and Safety of Losartan/HCTZ Combination as Compared to Losartan Monotherapy in Pediatric Patients With Essential Hypertension
Brief Title: A Study of Losartan Compared to Losartan/HCTZ in Pediatric Patients With Hypertension (0954A-327)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Achieving site readiness and enrolling the trial within a reasonable time
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954A-327; 2007_502
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — hydrochlorothiazide, losartan drug combination; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Losartan 50 mg (Active Comparator): Losartan 50 mg tablet, oral, once daily for 4 weeks. Participant also will be co-administered placebo for losartan 50 mg/hydrochlorothiazide (HCTZ) 12.5 mg once daily for 4 weeks
  Interventions: Drug: losartan potassium; Drug: Placebo for Losartan/HCTZ
- Losartan 100 mg (Active Comparator): Losartan 100 mg tablet, oral, once daily for 4 weeks. Participant also will be co-administered placebo for losartan 100 mg/hydrochlorothiazide (HCTZ) 12.5 mg once daily for 4 weeks
  Interventions: Drug: losartan potassium; Drug: Placebo for Losartan/HCTZ
- Losartan 50 mg/HCTZ 12.5 mg (Experimental): Losartan 50 mg/hydrochlorothiazide (HCTZ) 12.5 mg tablet, oral, once daily for 4 weeks. Participant also will be co-administered placebo for losartan 50 mg once daily for 4 weeks
  Interventions: Drug: hydrochlorothiazide (+) losartan potassium; Drug: Placebo for Losartan
- Losartan 100 mg/HCTZ 12.5 mg (Experimental): Losartan 100 mg/hydrochlorothiazide (HCTZ) 12.5 mg tablet, oral, once daily for 4 weeks. Participant also will be co-administered placebo for losartan 100 mg once daily for 4 weeks
  Interventions: Drug: hydrochlorothiazide (+) losartan potassium; Drug: Placebo for Losartan

INTERVENTIONS:
Drug: hydrochlorothiazide (+) losartan potassium — losartan/hydrochlorothiazide 12.5mg tablet po qd; for a 4 week study period.
  Other Names: MK0954A
  Arms: Losartan 100 mg/HCTZ 12.5 mg; Losartan 50 mg/HCTZ 12.5 mg
Drug: losartan potassium — Losartan 50mg titrating up to Losartan 100mg tablet po qd; for a 4 week study period
  Other Names: MK0954
  Arms: Losartan 100 mg; Losartan 50 mg
Drug: Placebo for Losartan
  Arms: Losartan 100 mg/HCTZ 12.5 mg; Losartan 50 mg/HCTZ 12.5 mg
Drug: Placebo for Losartan/HCTZ — losartan/hydrochlorothiazide 12.5mg Pbo tablet po qd; for a 4 week study period.
  Arms: Losartan 100 mg; Losartan 50 mg

SUMMARY:
The purpose of this study is to test the safety and effectiveness of Losartan as compared to Losartan/HCTZ in pediatric patients (6 to 17 years) with high blood pressure.

DETAILED DESCRIPTION:
Participants who meet eligibility requirements will enter the single-blind Filter Period. Participants with either sitting systolic blood pressure (SiSBP) or sitting diastolic blood pressure (SiDBP) >=95th percentile for gender/age/height will be administered either losartan 25 mg or losartan 50 mg depending on body weight (<50 kg and >=50 kg, respectively). After 3 weeks, if SiSBP or SiDBP is >=95th percentile, participants will titrate to either losartan 50 mg or 100 mg according to weight. Participants with both SiSBP and SiDBP <95th percentile will be excluded from the study. After an additional 3 weeks, participants whose blood pressure (either SiSBP or SiDBP) remains >=95th percentile will then enter the double-blind phase. Participants who meet all entry criteria will be randomized in a 1:1 fashion to either losartan or losartan/hydrochlorothiazide (HCTZ) for 4 weeks and will be stratified according to body weight (<50 kg and >=50 kg). Participants whose weight is <50 kg will be randomized to losartan 50 mg or losartan50 mg/HCTZ 12.5 mg. Participants weighing >=50 kg will be randomized to losartan 100 mg or losartan/HCTZ 100 mg/12.5 mg. At the end of double-blind treatment, participants may enter a 20-week double-blind extension and will continue on their randomized therapy with losartan or losartan/HCTZ.

40 participants were enrolled and screened; the trial was terminated before any participants were randomized into the double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male/female and 6 to 17 years of age at the time of study with hypertension (high blood pressure)
* Patient is able to swallow tablets
* Females of child bearing potential must use acceptable contraception throughout the trial

Exclusion Criteria:

* Patient has a history of heart, metabolic or kidney disease
* Patient has a history of known heart, lung, liver and other body system disorders
* Patient is pregnant or nursing
* Patient has participated in another clinical trial within the last 28 days

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2007-05-24 (Actual); Primary Completion 2007-10-22 (Actual); Study Completion 2007-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was discontinued early due to limited availability of sites and readiness of sites to enroll participants within the predefined time. Although some participants were screened and entered Filter Period, none were randomly assigned to a treatment arm and none entered double-blind treatment period.
Pre-assignment Details: Enrolled participants entered screening. If initial criteria were met, eligible participants were separated into 2 strata based on weight and administered either 25-50mg or 50-100mg Losartan during Filter Period. Participant's whose blood pressure did not respond were eligible to be randomly assigned to the Treatment period of the study.
Groups:
- All Enrolled: Participants who met initial screening criteria for inclusion in study and were enrolled in the study.
- Losartan 25 Mg-50 mg (Filter Period): Participants <50 kg; Administered Losartan 25 mg, oral, once daily for 3 weeks, then Losartan 50 mg for 3 weeks
- Losartan 50 Mg-100 mg (Filter Period): Participants >=50 kg; Administered Losartan 50mg, oral, once daily for 3 weeks, then Losartan 100 mg for 3 weeks
Period: Screening
Arm/Group | All Enrolled | Losartan 25 Mg-50 mg (Filter Period) | Losartan 50 Mg-100 mg (Filter Period)
Started | 40 | 0 | 0
Completed | 19 | 0 | 0
Not Completed | 21 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Screen Failure | 4 | 0 | 0
Not completed — Study Terminated by Sponsor | 15 | 0 | 0
Period: Filter Period
Arm/Group | All Enrolled | Losartan 25 Mg-50 mg (Filter Period) | Losartan 50 Mg-100 mg (Filter Period)
Started | 0 | 4 (The study was discontinued early; no participant entered treatment period) | 15 (The study was discontinued early; no participant entered treatment period)
Completed | 0 | 0 | 0
Not Completed | 0 | 4 | 15
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Screen Failure | 0 | 3 | 4
Not completed — Study terminated by Sponsor | 0 | 1 | 10

BASELINE CHARACTERISTICS:
Population: All enrolled population which included all participants who provided consent and entered screening period of study.
Arm/Group | All Enrolled
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.7 (2.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Sitting Trough Systolic Blood Pressure (SiSBP) at Week 4 of Double-blind Treatment Period
Time Frame: Baseline and Week 4
Population: Full Analysis Set (FAS) Population, defined as all participants who were randomly assigned to a treatment arm for double-blind treatment period of study. This analysis was not done. The study was terminated before any participants were randomized to a treatment arm.
Arm/Group | Losartan 50 mg | Losartan 100 mg | Losartan 50 mg/HCTZ 12.5 mg | Losartan 100 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Experience an Adverse Event During Double-blind Treatment Phase of Study
Time Frame: up to 4 weeks
Population: All Participants as Treated (APaT) Population, defined as participants who were randomly assigned to a treatment arm and who received at least 1 dose of study therapy. Study terminated early; no participant entered treatment period of study.
Arm/Group | Losartan 50 mg | Losartan 100 mg | Losartan 50 mg/HCTZ 12.5 mg | Losartan 100 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Had Study Drug Discontinued Due to an Adverse Event During Double-blind Treatment Phase of Study
Time Frame: up to 4 weeks
Population: as for outcome 2
Arm/Group | Losartan 50 mg | Losartan 100 mg | Losartan 50 mg/HCTZ 12.5 mg | Losartan 100 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Sitting Trough Diastolic Blood Pressure (SiDBP) at Week 4 of Double-blind Treatment Period
Time Frame: Baseline and Week 4
Population: as for outcome 1
Arm/Group | Losartan 50 mg | Losartan 100 mg | Losartan 50 mg/HCTZ 12.5 mg | Losartan 100 mg/HCTZ 12.5 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 6 weeks (Filter period)
Description: Adverse events are reported for the 19 participants who were enrolled and entered the Filter Period. No participants entered the planned double-blind treatment period of this study.
Arm/Group | Losartan 25 Mg-50 mg (Filter Period) | Losartan 50 Mg-100 mg (Filter Period)
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/15
Other Adverse Events (participants affected / at risk) | 1/4 | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan 25 Mg-50 mg (Filter Period) (N=4) | Losartan 50 Mg-100 mg (Filter Period) (N=15)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was discontinued early (during screening) due to limited availability of sites and readiness of sites to enroll participants within the predefined time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.